CLINICAL TRIAL: NCT05280665
Title: The Impact of Specialization on Clinical Outcomes in Gastric Cancer Surgery
Brief Title: Specialization in Gastric Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Ali GUNER, Professor, MD, Karadeniz Technical University
Other Study IDs: GastCaSpec
Record Dates: First submitted 2022-02-22; First posted 2022-03-15 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Stomach Neoplasms; Gastric Cancer
Keywords: Specialization; Postoperative Complications; Morbidity; Gastrectomy; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The non-specialized group: Patients who were operated by a non-specialized surgeon. Non-specialized surgeons were defined as general surgeon who does not have the characteristics of a specialized gastric cancer surgeon.
  The non-specialized group will be divided into two subgroups (high-volume vs low-volume) for further analysis.
- The specialized group: Patients who were operated by a specialized gastric cancer surgeon. Specialized gastric cancer surgeons were defined as surgeons who meet all of the criteria for a specialized gastric cancer surgeon.
  * Who had undergone professional training in gastric cancer surgery in specialized gastric cancer centers (in Japan or Korea),
  * Who identified themselves as primarily gastric surgeons during the study period
  * Whose annual gastric cancer surgery volume is more than 21
  Interventions: Other: Specialization

INTERVENTIONS:
Other: Specialization — * Who had undergone professional training in gastric cancer surgery in specialized gastric cancer centers (in Japan or Korea),
  * Who identified themselves as primarily gastric surgeons during the study period
  * Whose annual gastric cancer surgery volume is more than 21
  Other Names: Gastric cancer surgery
  Groups: The specialized group

SUMMARY:
Specialization is having competent and effective knowledge on a subject, and the tendency towards specialization is increasing due to the fact that it increases the success in the follow-up and treatment process of diseases. It has been observed that specialization in cancer surgery provides significant improvement in clinical outcomes in recent years. In this study, the effect of specialization in gastric cancer surgery on clinical outcomes is being investigated.

DETAILED DESCRIPTION:
Specialization is having sufficient and effective knowledge on a subject. Today, in the medical world, specialization is defined as having competent knowledge on a disease, and in recent years, the benefit of specialization has begun to be emphasized. Initially, it was defined as a branching and over the years, internal and surgical departments were divided into sub-areas. In surgical sciences, these fields are determined as traumatology, breast-endocrine surgery and gastrointestinal system surgery. This branching has brought a different perspective and approach to diseases and has made it possible to be more effective in the management of diseases. In recent years, a specialization approach on diseases and organ systems has developed within these branches. In surgery, surgeons specialized on many organs such as pancreatic surgery, colorectal surgery, gastric surgery, breast surgery, ovarian surgery have increased the efficiency in the management of diseases and the survival and disease-free survival rates of the patients have increased, and the postoperative morbidity and mortality rates have decreased.

Gastric cancer is one of the most common malignant cancers. It is the fifth most common cause of cancer-related death worldwide. Despite advances in diagnosis and treatment methods, patients may still be diagnosed late, and patients still have a poor prognosis due to the biology of gastric cancer. Even in properly treated patients, five-year survival rates are around 20-30%. With the development of surgical techniques and disease management, clinical outcomes of the disease have improved and mortality has been reduced. In the studies, the definition of gastric surgeon was created and it was determined that the mortality decreased proportionally with the increase in the patient volume of the surgeon. In gastric cancer surgery, there are mostly studies on the number of surgeon patients and the number of hospital patients. Post-hoc analysis of hospital volume on patients included in the CRITICS study showed a 13.1% increase in survival in high-volume hospitals compared to low-volume hospitals. The number of annual resections ≥21 was determined as the definition of high-volume hospital. In addition, it was determined that there was a decrease in mortality as the number of annual cases increased in high-volume hospitals. In another study, it was seen that there was an improvement in the mortality of medium and high volume hospitals compared to low volume hospitals. The majority of studies in gastric cancer surgery have focused on hospital volume and surgeon volume. There are no data on the specialization of the surgeon other than a study based in Japan.

In this study, it was aimed to evaluate the effect of specialization in gastric cancer surgery on short- and long-term clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* cStage I/II/III gastric cancer
* Histologically proven gastric adenocarcinoma
* Underwent surgery with curative intent

Exclusion Criteria:

* Under 18 years old
* Patients with non-adenocarcinoma diagnosis
* Emergency surgeries
* The need for a thoracic approach
* Patients with a history of non-gastric cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical stage 1-3 gastric adenocarcinoma undergoing surgical treatment for curative purposes
Sampling Method: Probability Sample
Enrollment: 537 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30 days after the operation (postoperative hospital stay ≤ 30 days) or operation to first discharge from hospital (postoperative hospital stay > 30 days)
  Death from any cause within 30 days after surgery or at any time if not discharged from hospital

SECONDARY OUTCOMES:
90-day mortality | 90 days after the operation (postoperative hospital stay ≤ 90 days) or operation to first discharge from hospital (postoperative hospital stay > 90 days)
  Death from any cause within 90 days after surgery or at any time if not discharged from hospital
Postoperative complication rate | Within 30 days after the operation
  Any complications (graded by the Clavien-Dindo classification) occurred in the postoperative period
Postoperative major complication rate | Within 30 days after the operation
  ≥grade-III Clavien-Dindo complications occurred in the postoperative period
Readmission | Within 30 days after the operation
  Readmission requiring re-hospitalization for any complications after discharge
3-year overall survival | 3 years after surgery
  Death from any cause is defined as an event.
3-year recurrence-free survival | 3 years after surgery
  Death from any cause or the recurrence of gastric cancer are an event.
Hospital stay | From the date of surgery until the date of hospital discharge, assessed up to 90 days after the operation
  Duration of postoperative hospital stays

OTHER OUTCOMES:
Failure-to-cure | Within 30 days after the operation
  futile surgery due to intraoperative distant metastasis/irresectability, OR microscopically or macroscopically incomplete resection OR 30-day mortality
Neoadjuvant treatment usage | Within the three months before surgery
  Neoadjuvant treatment usage rates in patients undergoing surgical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ali Guner, MD, Principal Investigator — Karadeniz Technical University Faculty of Medicine
Locations (1):
- Karadeniz Technical University, Faculty of Medicine, Farabi Hospital, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
With a reasonable request, we are open to share IPD.

REFERENCES:
- [Background] Liang Y, Wu L, Wang X, Ding X, Liang H. The positive impact of surgeon specialization on survival for gastric cancer patients after surgery with curative intent. Gastric Cancer. 2015 Oct;18(4):859-67. doi: 10.1007/s10120-014-0436-1. Epub 2014 Oct 15. PMID 25315086
- [Background] Bachmann MO, Alderson D, Edwards D, Wotton S, Bedford C, Peters TJ, Harvey IM. Cohort study in South and West England of the influence of specialization on the management and outcome of patients with oesophageal and gastric cancers. Br J Surg. 2002 Jul;89(7):914-22. doi: 10.1046/j.1365-2168.2002.02135.x. PMID 12081743
- [Background] Claassen YHM, van Amelsfoort RM, Hartgrink HH, Dikken JL, de Steur WO, van Sandick JW, van Grieken NCT, Cats A, Boot H, Trip AK, Jansen EPM, Kranenbarg EM, Braak JPBM, Putter H, van Berge Henegouwen MI, Verheij M, van de Velde CJH. Effect of Hospital Volume With Respect to Performing Gastric Cancer Resection on Recurrence and Survival: Results From the CRITICS Trial. Ann Surg. 2019 Dec;270(6):1096-1102. doi: 10.1097/SLA.0000000000002940. PMID 29995679
- [Background] Callahan MA, Christos PJ, Gold HT, Mushlin AI, Daly JM. Influence of surgical subspecialty training on in-hospital mortality for gastrectomy and colectomy patients. Ann Surg. 2003 Oct;238(4):629-36; discussion 636-9. doi: 10.1097/01.sla.0000089855.96280.4a. PMID 14530734